CLINICAL TRIAL: NCT01857193
Title: A Phase Ib Trial of LEE011 in Combination With Everolimus (RAD001) and Exemestane in the Treatment of Postmenopausal Women With Hormone Receptor Positive, HER2 Negative Locally Advanced or Metastatic Breast Cancer
Brief Title: Phase Ib Trial of LEE011 With Everolimus (RAD001) and Exemestane in the Treatment of Hormone Receptor Positive HER2 Negative Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011X2106
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: Open label; dose escalation; ER+; LEE011; CDK4/6; everolimus; advanced breast cancer; mTOR; HR positive; HER2 negative
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; exemestane; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- L-R-E arm (Experimental): Participants who took ribociclib (LEE011), everolimus (RAD001) and exemestane triple combination
  Interventions: Drug: ribociclib (LEE011); Drug: Exemestane; Drug: Everolimus (RAD001)
- L-E arm (Experimental): Participants who ribociclib (LEE011) and exemestane double combination
  Interventions: Drug: ribociclib (LEE011); Drug: Exemestane

INTERVENTIONS:
Drug: ribociclib (LEE011) — LEE011 is taken orally once per day for 21 days of each 28 day cycle. LEE011 comes in 50 mg and 200 mg capsules.
  Other Names: LEE011
Drug: Exemestane — Exemestane is taken orally once per day. Exemestane comes in 25 mg tablets.
Drug: Everolimus (RAD001) — Everolimus is taken orally once per day. Everolimus comes in 1 mg, 2.5 mg, 5mg, and 7.5 mg tablets
  Other Names: RAD001
  Arms: L-R-E arm

SUMMARY:
Dose Escalation part of the study: To estimate the MTD(s) and/ or RP2D of LEE011 in combination with everolimus + exemestane, and LEE011 in combination with exemestane, and to characterize the safety and tolerability of the combinations of everolimus + exemestane + LEE011 and LEE011 + exemestane in patients with ER+ HER2- advanced breast cancer

Dose Expansion part of the study: To characterize the safety and tolerability of the triplet combination of LEE011 + everolimus + exemestane in patients naïve or refractory to CDK4/6 inhibitor based therapy, and the safety and tolerability of the doublet combination of LEE011 + exemestane in patients refractory to CDK4/6 inhibitor based therapy (except patients treated with prior LEE011 are not allowed in Group 3).

DETAILED DESCRIPTION:
The primary purpose of the phase Ib part of this study is to determine the maximum tolerated dose(s) (MTD(s)) and/or recommended phase II dose (RP2D) of LEE011 + everolimus + exemestane in patients with ER+ Her2- advanced breast cancer. This part of the study will also assess safety, tolerability, and PK of the LEE011 + exemestane, LEE011 + everolimus + exemestane combinations.

The Dose Expansion part of the study will evaluate the triple combination of LEE011 + everolimus + exemestane and the double combination of LEE011 + exemestane for safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥ 18 years of age) with metastatic or locally advanced breast cancer
* Histological or cytological confirmation of ER+ breast cancer in dose escalation and HR+ breast cancer in dose expansion
* A representative tumor specimen must be available for molecular testing.
* Postmenopausal women. Postmenopausal status is defined either by:
* Age ≥ 18 with prior bilateral oophorectomy
* Age ≥ 60 years
* Age <60 years with amenorrhea for at least 12 months and both follicle-stimulating hormone (FSH) and estradiol levels are in postmenopausal range (according to the local laboratory)
* Recurrence while on, or within 12 months of end of adjuvant treatment with letrozole or anastrozole, or
* Progression while on, or within one month of end of letrozole or anastrozole treatment for locally advanced or metastatic breast cancer.
* Patients must have:

  * Measurable disease*: At least one lesion that can be accurately measured in at least one dimension ≥ 20 mm with conventional imaging techniques or ≥ 10 mm with spiral CT or MRI or
  * Bone lesions: lytic or mixed (lytic + sclerotic) in the absence of measurable disease as defined above.
* ECOG Performance Status 0-1.
* Fasting serum cholesterol ≤ 300 mg/dl or 7.75 mmol/L and fasting triglycerides ≤ 2.5 × ULN. In case one or both of these thresholds are exceeded, the patient can only be included after initiation of statin therapy and when the above mentioned values have been achieved
* Standard 12-lead ECG values defined as the mean of the triplicate ECGs and assessed by the central laboratory.

  * QTcF interval at screening < 450 msec (using Fridericia's correction).
  * Resting heart rate 50-90 bpm

Exclusion Criteria:

* HER2-overexpressing patients by local laboratory testing (IHC 3+ staining or in situ hybridization positive).
* Patients who received more than one chemotherapy line for advanced breast cancer.
* Previous treatment with exemestane or mTOR inhibitors* (Note:

Patients with disease refractory to prior LEE011 are excluded for dose expansion Group 3 only).

* History of brain or other CNS metastases.
* Clinically significant, uncontrolled heart disease and/or recent cardiac repolarization abnormality including any of the following:
* History of myocardial infarction (MI), angina pectoris, symptomatic pericarditis, or coronary artery bypass graft (CABG) within 6 months prior to study entry
* Documented cardiomyopathy
* Left ventricular ejection fraction (LVEF) < 50% as determined by Multiple Gated acquisition scan (MUGA) or echocardiogram (ECHO)
* Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, and etc.
* Clinically significant cardiac arrhythmias, complete left bundle branch block, high-grade AV block
* Systolic Blood Pressure (SBP) >160 or <90 mmHg
* Patients who are currently receiving treatment with agents that are known to cause QTc prolongation in humans
* Patients who are currently receiving treatment (within 7 days prior to starting study treatment) with strong and moderate inhibitors or inducers of CYP3A4/5, substrates of CYP3A4/5 with a narrow therapeutic index or Herbal preparations/medications (Refer to Section 6.4 and Appendix 3)

Inclusion Criteria Exceptions for Phase Ib Dose Expansion patients:

Dose Expansion part of the study has 3 groups, following are the Inclusion Criteria exceptions for these 3 groups

1. Group 1 - Patients must not have received prior treatment with any CDK4/6 inhibitors
2. Group 2 - Patients must have disease progression while on or within one month after CDK4/6 inhibitor based therapy
3. Group 3 - Patients must have disease progression while on or within one month after CDK4/6 inhibitor based therapy (except those patients who received prior LEE011 based therapy).

Other protocol-defined Inclusion/Exclusion may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-09-06 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Incidence of Dose Limiting Toxicity (DLT) | At the end of Cycle 1 (each cycle is 28 days)
  DLT is defined as treatment-related toxicity (classified according Common Toxicity Criteria for Adverse Events (CTCAE) Version 4) occurring during the first 28 treatment days and meeting specific protocol-predefined criteria.
Dose Expansion: Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Approximately 4.5 years after FPFV
  Adverse events were collected for approximately 4.5 years for dose expansion including the 30 days safety follow-up period.

SECONDARY OUTCOMES:
Dose Escalation: Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Approximately 6.5 years after FPFV
  Adverse events were collected for approximately 6.5 years for dose escalation including the 30 days safety follow-up period.
Dose Escalation and Expansion: Overall Response Rate (ORR) | Approximately 6.5 years for Dose Escalation and 4.5 years for Dose Espansion after FPFV
  Overall Response Rate (ORR) is defined as the proportion of participants with a best overall response of complete response or partial response.
Dose Escalation and Expansion: Disease Control Rate (DCR) | Approximately 6.5 years for Dose Escalation and 4.5 years for Dose expansion after FPFV
  Disease Control Rate (DCR) is the proportion of patients with a best overall response of Complete Response or Partial Response or Stable Disease.
Dose Escalation and Expansion: Clinical Benefit Rate (CBR) | Approximately 6.5 years for Dose Escalation and 4.5 years for Dose Espansion after FPFV
  Clinical Benefit Rate (CBR) is the Complete Response, Partial Response, or Stable Disease lasting 24 weeks or longer
Dose Expansion: Duration of Response (DOR) | Approximately 4.5 years for dose expansion after FPFV
  Duration of Response (DOR) is calculated as the time from the date of first documented response (complete response (CR) or partial response (PR)) to the first documented date of progression or death due to underlying cancer. The DOR is not applicable as none of the patients in the expansion treatment groups (triplet treatment naive, triplet treatment refractory and doublet treatment refractory) had a CR or PR
Dose Expansion: Progression Free Survival (PFS) | Approximately 4.5 years after FPFV
  Progression Free Survival (PFS) is defined as the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment.
Dose Escalation: Pharmacokinetics (PK) parameter: AUC0-24h at Day 1 of Cycle 1 | 6 Cycles of treatment (28 day cycles): Cycle 1 Day 1
  AUC0-24h is the area under the drug concentration-time curve during a dosing interval (mass x time x volume-1).
Dose Escalation: Pharmacokinetics (PK) parameter: AUC0-24h at at Day 15 of Cycle 1 | 6 Cycles of treatment (28 day cycles): Cycle 1 Day 15
  AUC0-24h is the area under the drug concentration-time curve during a dosing interval (mass x time x volume-1).
Dose Escalation: Pharmacokinetics (PK) parameter: Cmax at Day 1 of Cycle 1 | 6 Cycles of treatment (28 day cycles): Cycle 1 Day 1
  Cmax is the maximum observed drug concentration after drug administration (mass x volume-1).
Dose Escalation: Pharmacokinetics (PK) parameter: Cmax at Day 15 of Cycle 1 | 6 Cycles of treatment (28 day cycles): Cycle 1 Day 15
  Cmax is the maximum observed drug concentration after drug administration (mass x volume-1).
Dose Escalation: Pharmacokinetics (PK) parameter: Tmax at Day 1 of Cycle 1 | 6 Cycles of treatment (28 day cycles): Cycle 1 Day 1
  Tmax is the time to reach maximum plasma/blood/serum drug concentration (time).
Dose Escalation: Pharmacokinetics (PK) parameter: Tmax at Day 15 of Cycle 1 | 6 Cycles of treatment (28 day cycles): Cycle 15 Day 1
  Tmax is the time to reach maximum plasma/blood/serum drug concentration (time).
Dose Escalation: Pharmacokinetics (PK) parameter: Racc at Day 15 of Cycle 1 | 6 Cycles of treatment (28 day cycles): Cycle 15 Day 1
  Racc is the accumulation ratio calculated as AUCtau,ss / AUCtau,sd

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (8):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Sylvester Comprehensive Cancer Center Main Center, Miami, Florida
  - Massachusetts General Hospital Onc Dept, Boston, Massachusetts
  - Karmanos Cancer Institute Dept of Onc, Detroit, Michigan
  - Memorial Sloan Kettering Oncology Dept., New York, New York
  - Oregon Health and Science University SC-5, Portland, Oregon
  - University of Texas MD Anderson Cancer Center Onc Dept, Houston, Texas
  - Northwest Medical Specialties, Tacoma, Washington
- Novartis Investigative Site, Wilrijk, Belgium
- Novartis Investigative Site, Saint-Herblain, France
- Novartis Investigative Site, Hong Kong, Hong Kong
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CLEE011X2106 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17815